CLINICAL TRIAL: NCT05654844
Title: Comparison of Linear And Angular Measurements in Mandibular Symphyseal Region Using Lateral Cephalometric and Cone Beam CT Images
Brief Title: Comparison of Lateral Cephalometric and Cone Beam CT Measurements in Mandibular Symphysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Erinc Onem, DDS, PhD, Professor, Ege University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: comparison of LC and CBCT
Record Dates: First submitted 2022-12-08; First posted 2022-12-16 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Measurements in Mandibular Symphysis
Keywords: mandibular symphysis; lateral cephalometry; cone beam CT

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Digital Lateral Cephalometry (Other): Patients justifying the indication for LC and CBCT exposure
  Interventions: Radiation: LC images; Radiation: CBCT images

INTERVENTIONS:
Radiation: LC images — Angular and Linear Measurements were compared in mandibular symphysis region using the LC images
Radiation: CBCT images — Angular and Linear Measurements were compared in mandibular symphysis region using the CBCT images

SUMMARY:
The goal of this clinical trial is to compare the linear and angular measurements of the mandibular symphyseal region using lateral cephalometric (LC) and cone beam computed tomography (CBCT) images. The main question it aims to answer are:

Is there a significant difference in measurements on lateral cephalometric and cone beam CT? Measurements were made by 3 radiologists, and the intra-class correlation coefficient (ICC) was used to measure interobserver reliability.

DETAILED DESCRIPTION:
The aim of the study is to compare the linear and angular measurements of the mandibular symphyseal region using lateral cephalometric (LC) and cone beam computed tomography (CBCT) images. One hundred patients justifying both LC and CBCT exposures were included. Both lateral cephalometric and CBCT images of the patients were used for angular and linear measurements. Angular measurements included vestibular-concavity, lingual- and tooth-inclination angles. Vestibular and lingual cortical bone and total bone thickness measurements were obtained for the comparison of linear measurements. Three radiologists performed the measurements on 200 images. Comparison of the measurements and the imaging methods were done using paired- and Wilcoxon t-tests. Inter-observer reliability was evaluated with the intra-class correlation coefficient (ICC).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 25 to 40 years with lateral cephalometric and CBCT exposure indication for various reasons and/or dental procedures.

Exclusion Criteria:

* Patients under 25 and above 40 years of age, with more than single missing mandibular anterior teeth, with implants and/or metal restorations in the mandibular anterior region that may disrupt image quality and thus measurements, prominent asymmetry of the mandibular anterior region, having orthodontic appliances, temporomandibular joint and/or muscle disorders and history of trauma were excluded from the study.

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2020-12-29 (Actual); Study Completion 2020-12-29 (Actual)

PRIMARY OUTCOMES:
Angular measurement-1 | 4 weeks
  Vestibular Concavity Angle (VCA) measurements had completed by 3 investigator on both images
Angular measurement-2 | 4 weeks
  Tooth Inclination Angle (TIA) measurements had completed by 3 investigator on both images
Angular measurement-3 | 4 weeks
  Lingual Inclination Angle (LIA) measurements had completed by 3 investigator on both images
Linear measurement-1 | 4 weeks
  Vestibular cortical bone thickness measurements had completed by 3 investigator on both images
Linear measurement-2 | 4 weeks
  Lingual cortical bone thickness (LCT) had completed by 3 investigator on both images
Linear measurement-3 | 4 weeks
  Total bone thickness (TBT) measurements had completed by 3 investigator on both images

CONTACTS AND LOCATIONS:
Overall Officials: Erinç Onem, Prof, Study Director — Academician in Ege University; Oguzhan Baydar, MSD, Principal Investigator — Master of Science in Dentistry in Ege University; B. Guniz Baksi, Prof, Study Chair — Academician in Ege University
Locations (1):
- Ege University, School of Dentistry, Izmir, Bornova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Houston WJ, Maher RE, McElroy D, Sherriff M. Sources of error in measurements from cephalometric radiographs. Eur J Orthod. 1986 Aug;8(3):149-51. doi: 10.1093/ejo/8.3.149. No abstract available. PMID 3464438
- [Background] Rai S, Misra D, Misra A, Kidwai S, Bisla S, Jain A, Gangwal P. Evaluation of neurovascular anatomical variation in the anterior mandible in North Indian population: A CBCT assessment. J Oral Biol Craniofac Res. 2022 Sep-Oct;12(5):505-511. doi: 10.1016/j.jobcr.2022.06.005. Epub 2022 Jun 17. PMID 35783918
- [Background] Kumar V, Ludlow JB, Mol A, Cevidanes L. Comparison of conventional and cone beam CT synthesized cephalograms. Dentomaxillofac Radiol. 2007 Jul;36(5):263-9. doi: 10.1259/dmfr/98032356. PMID 17586852